CLINICAL TRIAL: NCT02192866
Title: Blood Samples for the Study of Peanut, Tree Nut and Other Food Allergies
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 13-2102; UL1TR001082 (NIH)
Record Dates: First submitted 2014-02-24; First posted 2014-07-17 (Estimated); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Peanut Allergies; Tree Nut Allergies; Other Food Allergies
MeSH Terms: conditions — Peanut Hypersensitivity; Nut Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Peanut allergic: No intervention(s) to be administered.
- Other food allergic: No intervention(s) to be administered.
- Controls: No intervention(s) to be administered.

SUMMARY:
Food allergies are now a major problem. These experiments involve getting blood from people with food allergies and from people without food allergies. The blood collected will be used to answer questions and find information about peanut and other food allergies.

Samples will come from:

* People signed up by the investigators at the University of Colorado Denver
* University of North Carolina, Massachusetts General Hospital, Children's Hospital of Colorado and the Immune Tolerance Network (Benaroya Research Institute) where people have been treated for peanut allergies
* University of North Carolina, Massachusetts General Hospital, National Jewish Health and The Children's Hospital in Denver where people have taken part or will take part in clinically indicated oral food challenges.

Blood and health histories from the University of North Carolina, Massachusetts General Hospital, National Jewish Health, The Children's Hospital and the Immune Tolerance Network will not have personal information linked.

The specific aims of this experiment are:

1. Come up with a lab test that will predict how bad an allergic reaction will be to peanuts.
2. Find out what part of a peanut causes allergic reactions.
3. Come up with preventions that can block peanut allergies.
4. Find the strongest proteins in walnuts.

DETAILED DESCRIPTION:
Overview: This is a protocol for obtaining serum, plasma, and cells from subjects with specific food allergies and from controls to be used in studies of peanut and other allergens. We are only asking the CTRC for help with drawing blood, separating serum, labeling tubes and to aliquot the serum. In addition, we will receive de-identified serum and plasma from other institutions and de-identified cord blood from the University of Colorado Denver Cord Blood bank.

The previous version of this application was COMIRB protocol 09-0813. This was last updated 03-03-2016. Much of the work outlined in protocol 09-0813 was completed and a manuscript is under review. This protocol is still only for the purpose of drawing blood and obtaining clinical histories. As such the risks and benefits in the informed consent have not changed.

Based on new NIH funding (RO3 AI 164349; started 7-09-21) and RO1-AI165866 (9th %-tile; scheduled to begin 09-01-21), the project now includes 5 specific aims (Aims #1-5). Aims 1 & 2 are part of an R21 funded project (R21 AI135397; 11/16/2018-10/31/2020; extended until 10/31/2021 without additional funds) to Dr. Dreskin. Aims 3 & 4 are part of an R21 funded project (R21 AI137881; 11/28/2018-10/31/2020; extended until 10/31/2021 without additional funds) to Dr. Chen (Dr. Dreskin is Co-PI). These proposals are highly complementary and each only needs access to blood samples. Dr. Dreskin's proposal consists of in vitro experiments to test IgE binding to novel peptides. Dr. Chen's proposal uses human serum or plasma as a source of IgE with which to identify and characterize mimotopes for murine studies. Aim 5 is an exploratory aim to obtain preliminary data for an RO1 to be submitted in 2019. For all of these projects, the only experiments that involve human materials are ex vivo assays of basophil activation, in vitro assays of IgE binding and generation of humanized mice using de-identified cord blood that will otherwise be discarded. There are no therapeutic interventions for human subjects.

ELIGIBILITY:
Inclusion Criteria:

This protocol is to draw blood for a variety of related studies of food allergy. For this reason, we will list each group of subjects and the inclusion criteria for that group.

1. De-identified sera or plasma from patients who have undergone Oral ImmunoTherapy (OIT) for peanut allergy. These samples already exist.

   * Inclusion criteria:

     1. patients have been enrolled in a controlled trial of OIT for peanuts, and had at least one oral challenge.
     2. Age 1-75.
2. De-identified samples from patients who are undergoing clinically indicated food challenges for peanut allergy.

   * Inclusion criteria:

     1. concern regarding possible allergy to peanuts,
     2. age 1-75,
     3. plan to undergo a clinically indicated challenge with peanuts.
3. Patients with peanut allergy.

   * Inclusion criteria:

     1. excellent history of a systemic reaction to peanuts,
     2. age 6-75.
4. Patients with other food allergies (especially tree nuts).

   * Inclusion criteria:

     1. excellent history of a systemic reaction to tree nuts or other foods,
     2. age 6-75.
5. Normal controls.

   * Inclusion criteria:

     1. no known food allergies,
     2. recent ingestion of peanuts without difficulty, and
     3. age 6-75.

Exclusion Criteria:

1. Any known significant medical or psychiatric diagnosis
2. Use of an investigational drug within 30 days
3. Use of omalizumab (anti-IgE; Xolair) within 6 months

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children who are allergic to peanuts and/or tree-nuts and individuals with no known food allergies.
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Identify which traits are associated with severe food allergy. | 1 day of single blood draw
  This is an observational study, to describe traits (identified through blood tests) associated with severe food allergy, particularly peanut allergy.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Dreskin, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado School of Medicine, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dreskin SC, Koppelman SJ, Andorf S, Nadeau KC, Kalra A, Braun W, Negi SS, Chen X, Schein CH. The importance of the 2S albumins for allergenicity and cross-reactivity of peanuts, tree nuts, and sesame seeds. J Allergy Clin Immunol. 2021 Apr;147(4):1154-1163. doi: 10.1016/j.jaci.2020.11.004. Epub 2020 Nov 18. PMID 33217410
- [Result] Hazebrouck S, Patil SU, Guillon B, Lahood N, Dreskin SC, Adel-Patient K, Bernard H. Immunodominant conformational and linear IgE epitopes lie in a single segment of Ara h 2. J Allergy Clin Immunol. 2022 Jul;150(1):131-139. doi: 10.1016/j.jaci.2021.12.796. Epub 2022 Feb 10. PMID 35150723
- [Result] Hazebrouck S, Canon N, Dreskin SC. The Effector Function of Allergens. Front Allergy. 2022 Feb 7;3:818732. doi: 10.3389/falgy.2022.818732. eCollection 2022. PMID 35386644
- [Result] Dreskin SC, Germinaro M, Reinhold D, Chen X, Vickery BP, Kulis M, Burks AW, Negi SS, Braun W, Chambliss JM, Eglite S, McNulty CMG. IgE binding to linear epitopes of Ara h 2 in peanut allergic preschool children undergoing oral Immunotherapy. Pediatr Allergy Immunol. 2019 Dec;30(8):817-823. doi: 10.1111/pai.13117. Epub 2019 Oct 21. PMID 31437325